CLINICAL TRIAL: NCT02426112
Title: Bronchopulmonary Function in Response to Azithromycin Treatment for Chronic Lung Disease in HIV-infected Children
Acronym: BREATHE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Biomedical Research and Training Institute, Zimbabwe (Other); Malawi-Liverpool-Wellcome Trust Clinical Research Programme (Other); University of Tromso (Other); University of Cape Town (Other); University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: QA698
Record Dates: First submitted 2015-04-21; First posted 2015-04-24 (Estimated); Last update posted 2019-10-09 (Actual); Status verified 2019-10

CONDITIONS: Chronic Lung Disease; HIV Infection
MeSH Terms: conditions — HIV Infections | interventions — Azithromycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Azithomycin (Active Comparator): Azithromycin tablets 250 mg, 30mg/kg/week by mouth, once a week for 12 months.
  * 10-20 kg: 250 mg
  * 20-29 kg: 500 mg
  * 30-39 kg: 750 mg
  * 40-49 kg: 1250 mg
  Interventions: Drug: Azithromycin
- Placebo (Placebo Comparator): Placebo tablets 250 mg, 30 mg/kg/week by mouth, once a week for 12 months.
  * 10-20 kg: 250 mg
  * 20-29 kg: 500 mg
  * 30-39 kg: 750 mg
  * 40-49 kg: 1250 mg
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Azithromycin
  Arms: Azithomycin
Drug: Placebo
  Arms: Placebo

SUMMARY:
Chronic pulmonary disease (CLD) is the most common manifestation of HIV/AIDS among children, accounting for more than 50% of HIV-associated mortality. Recently, a novel form of CLD, affecting more than 30% of African HIV-infected older children was described by Ferrand et al in Zimbabwe, high-resolution CT scanning findings showed predominantly small airways disease consistent with constrictive obliterative bronchiolitis (OB). . Azithromycin has anti-inflammatory activity and treatment of CLD with this agent may lead to suppression of generalized immune activation.

This specific aims of this project are to:

1. Primary objective: To investigate whether adjuvant treatment with azithromycin results in improvement in lung function in HIV-infected children with chronic lung disease, who are stable on antiretroviral therapy.
2. Secondary objectives:

   1. To investigate the intervention effect on mortality, exacerbations of lung disease, quality of life, morbidity.
   2. To investigate adverse events related to azithromycin treatment

In total, 400 children aged 6-16 years, living with HIV and diagnosed with CLD will be enrolled at Harare Children´s Hospital in Harare (Zimbabwe) and Queen Elizabeth Central Hospital in Blantyre (Malawi). These will receive weekly treatment with azithromycin or placebo during 12 months. Another 100 children (50 per site) living with HIV but with no CLD will be enrolled as a comparison group for laboratory sub-studies.

Lung function will be assess using spirometry and the Forced expiratory volume in the first minute (FEV1) will be the primary outcome. The mean change in FEV1 z-score levels will be compared between trial arms after 12 months of initiation of azithromycin treatment.

DETAILED DESCRIPTION:
Clinical Phase: III

Trial Design: Multi-site, individually randomised, double-blinded, placebo-controlled trial of weekly azithromycin for 12 months

Trial Participants: Children aged 6-16 years living with HIV and with diagnosis of chronic lung disease. Another 200 children living with HIV but with no chronic lung disease in a comparison arm.

Planned Sample Size: 400 cases and 100 in the comparison arm

Treatment duration: 12 months

Follow up duration: 18 months

Planned Trial Period: June 2016-September 2019

Objectives:

* Primary trial outcome: To investigate whether adjuvant treatment with azithromycin results in improvement in lung function in HIV-infected children with chronic lung disease, who are stable on antiretroviral therapy.
* Secondary trial outcomes:

.To investigate the intervention effect on mortality,exacerbations of lung disease, quality of life and morbidity..

.To investigate adverse events related to azithromycin treatment. .-Laboratory sub-studies .To determine the effect of azithromycin therapy on antimicrobial resistance in bacteria colonizing the respiratory tract.

.To investigate the diversity and composition of the respiratory microbiome in HIV-infected children with CLD.

.To investigate the diversity and composition of the gut microbiome in HIV-infected children with CLD.

.To investigate the effect of azithromycin on biomarkers of systemic inflammation in HIV-infected children with CLD.

.-Cardiac sub-study: .Describe the cardiac symptoms and echocardiograph findings of HIV-infected children with chronic lung disease.

.To investigate whether adjuvant treatment with azithromycin results in improvement in right-sided cardiac function and/or pulmonary hypertension in HIV-infected children with chronic lung disease.

Investigational Medicinal Product(s): Azithromycin and placebo.

Formulation:Tablets 250 mg

Dose: According to weight bands (30 mg/kg/week):

* 10-20 kg: 250 mg
* 20-29 kg: 500 mg
* 30-39 kg: 750 mg
* 40-49 kg: 1250 mg

Route of Administration:Oral

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of chronic lung disease (defined as FEV1 and/or FVC <80% predicted)
2. Age 6-19 years
3. Perinatally-acquired HIV infection the most likely source of transmission
4. On first or second-line ART for at least one year
5. HIV-1 viral load undetectable (as defined by each trial site)
6. A firm home address accessible for visiting and intending to remain there for 24 months
7. Willing to agree to participate in the study and to give samples of blood and sputum
8. HIV status disclosed to child for those aged older than 12 years

Exclusion Criteria:

1. Any condition (except HIV) that may prove fatal during the study period (e.g. malignancy, end-stage HIV disease or other conditions deemed likely fatal by the trial physician)
2. Diagnosis of active pulmonary TB
3. Infection with non-tuberculous mycobacteria (NTM)
4. Pregnant or breast-feeding
5. Condition likely to lead to lack of understanding of study procedures or to uncooperative behaviour e.g. neurocognitive disease, developmental delay or psychiatric illness
6. History of prolonged QTc syndrome or current or planned therapy with drugs likely to cause cardiac dysrhythmias
7. Abnormal ECG findings
8. Acute respiratory tract infection during enrolment (patients will be eligible once their acute infection is treated)
9. Creatinine clearance of <30mls/minute
10. ALT more than 2 times the upper limit of normal
11. No defined guardian/stable caregiver
12. No consent/assent from guardian/child

Ages: 6 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 347 (Actual)
Dates: Start 2016-06; Primary Completion 2018-09 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
Forced Expiratory Volume in one second z score (FEV1) | 12 months
  Change in FEV1after 12 months of initiation of therapy with azithromycin

SECONDARY OUTCOMES:
Forced Expiratory Volume in one second z score (FEV1) | 24 months
  Mean change in FEV1 24 months after treatment initiation with azithromycin
Time to death | 12 months
  Time to death 12 months after treatment initiation with azithromycin
Time to first acute exacerbation | 12 months
Number of hospitalizations | 12 and 24 months
Number of exacerbations | 12 and 24 months
Quality of life scores | 12 and 24 months
Mean change in weight-for-age z-score | 12 and 24 months
Number of mild, moderate and severe adverse events | 12 months
Number of Malaria episodes (Malawi only) | 12 months
Number of blood stream infections due to Salmonella typhi and non-typhi | 12 months
Number of gastroenteritis episodes | 12 months

OTHER OUTCOMES:
Macrolide resistance | 12 months
  Prevalence of colonization with macrolide (and multidrug-resistant) Streptococcus pneumoniae, Staphylococcus aureus and Haemophilus influenzae in the two trial arms at 12 months of initiation of treatment with azithromycin
Lung microbiome | baseline, 12 and 14 months
  Composition and diversity of the respiratory bacterial microbiome (determined by culture of clinically relevant organisms and sequencing of 16s rRNA gene amplicons)
Gut microbiome | baseline, 12 and 24 months
  Composition and diversity of the gut bacterial microbiome (determined by culture of clinically relevant organisms and sequencing of 16s rRNA gene amplicons
Inflammation biomarkers | baseline, 12 and 24 months
  Association between inflammation biomarker levels and FEV1
Cardiac dysfunction | Baseline
  prevalence of right sided cardiac dilatation and dysfunction
Cardiac dysfunction after treatment | 12 and 24 months
  Prevalence of right sided cardiac dilatation and dysfunction at 12 and 24 months of initiation of azithromycin therapy by intervention arm

CONTACTS AND LOCATIONS:
Overall Officials: Rashida Ferrand, Principal Investigator — London School of Hygiene and Tropical Medicine; Jon O Odland, Principal Investigator — University of Tromso
Locations (2):
- Malawi-Liverpool-Wellcome Trust Clinical Research Programme, Blantyre, Malawi
- Biomedical Research and Training Institute, Harare, Zimbabwe

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Mushunje PK, Sovershaeva E, Olwagen CP, Madhi S, Odland JO, Ferrand RA, Nicol MP, Abotsi RE, Dube FS. Weekly azithromycin for 48 weeks impacts nasopharyngeal microbial prevalence and Streptococcus pneumoniae serotypes in children with HIV-associated chronic lung disease. Sci Rep. 2025 Nov 7;15(1):39175. doi: 10.1038/s41598-025-23693-6. PMID 41203736
- [Derived] Madanhire T, McHugh G, Simms V, Ngwira L, Gonzalez-Martinez C, Semphere R, Moyo B, Calderwood C, Nicol M, Bandason T, Odland JO, Rehman AM, Ferrand RA. Longitudinal lung function trajectories in response to azithromycin therapy for chronic lung disease in children with HIV infection: a secondary analysis of the BREATHE trial. BMC Pulm Med. 2024 Jul 12;24(1):339. doi: 10.1186/s12890-024-03155-x. PMID 38997676
- [Derived] Mushunje PK, Dube FS, Olwagen C, Madhi S, Odland JO, Ferrand RA, Nicol MP, Abotsi RE; BREATHE study team. Characterization of bacterial and viral pathogens in the respiratory tract of children with HIV-associated chronic lung disease: a case-control study. BMC Infect Dis. 2024 Jun 26;24(1):637. doi: 10.1186/s12879-024-09540-5. PMID 38926682
- [Derived] Ngwira LG, Maheswaran H, Verstraete J, Petrou S, Niessen L, Smith SC. Psychometric performance of the Chichewa versions of the EQ-5D-Y-3L and EQ-5D-Y-5L among healthy and sick children and adolescents in Malawi. J Patient Rep Outcomes. 2023 Mar 9;7(1):22. doi: 10.1186/s41687-023-00560-4. PMID 36892714
- [Derived] Rehman AM, Simms V, McHugh G, Mujuru H, Ngwira LG, Semphere R, Moyo B, Bandason T, Odland JO, Ferrand RA. Adherence to additional medication for management of HIV-associated comorbidities among older children and adolescents taking antiretroviral therapy. PLoS One. 2022 Jun 15;17(6):e0269229. doi: 10.1371/journal.pone.0269229. eCollection 2022. PMID 35704559
- [Derived] Jackson C, Rehman AM, McHugh G, Gonzalez-Martinez C, Ngwira LG, Bandason T, Mujuru H, Odland JO, Corbett EL, Ferrand RA, Simms V. Risk factors for sustained virological non-suppression among children and adolescents living with HIV in Zimbabwe and Malawi: a secondary data analysis. BMC Pediatr. 2022 Jun 11;22(1):340. doi: 10.1186/s12887-022-03400-4. PMID 35690762
- [Derived] Ferrand RA, McHugh G, Rehman AM, Mujuru H, Simms V, Majonga ED, Nicol MP, Flaegstad T, Gutteberg TJ, Gonzalez-Martinez C, Corbett EL, Rowland-Jones SL, Kranzer K, Weiss HA, Odland JO; BREATHE Trial Group. Effect of Once-Weekly Azithromycin vs Placebo in Children With HIV-Associated Chronic Lung Disease: The BREATHE Randomized Clinical Trial. JAMA Netw Open. 2020 Dec 1;3(12):e2028484. doi: 10.1001/jamanetworkopen.2020.28484. PMID 33331916
- [Derived] Rehman AM, Ferrand R, Allen E, Simms V, McHugh G, Weiss HA. Exclusion of enrolled participants in randomised controlled trials: what to do with ineligible participants? BMJ Open. 2020 Dec 2;10(12):e039546. doi: 10.1136/bmjopen-2020-039546. PMID 33268410
- [Derived] McHugh G, Rehman AM, Simms V, Gonzalez-Martinez C, Bandason T, Dauya E, Moyo B, Mujuru H, Rylance J, Sovershaeva E, Weiss HA, Kranzer K, Odland J, Ferrand RA; BREATHE Clinical Trial Team. Chronic lung disease in children and adolescents with HIV: a case-control study. Trop Med Int Health. 2020 May;25(5):590-599. doi: 10.1111/tmi.13375. Epub 2020 Feb 10. PMID 31989731
- [Derived] Gonzalez-Martinez C, Kranzer K, McHugh G, Corbett EL, Mujuru H, Nicol MP, Rowland-Jones S, Rehman AM, Gutteberg TJ, Flaegstad T, Odland JO, Ferrand RA; BREATHE study team. Azithromycin versus placebo for the treatment of HIV-associated chronic lung disease in children and adolescents (BREATHE trial): study protocol for a randomised controlled trial. Trials. 2017 Dec 28;18(1):622. doi: 10.1186/s13063-017-2344-2. PMID 29282143